CLINICAL TRIAL: NCT03265951
Title: A Pilot, Randomized, Double-blind, Placebo Controlled, Trial of Ramelteon for CPAP Non-Adherent Veterans With PTSD and Complex Insomnia
Brief Title: Ramelteon for Complex Insomnia in Veterans With PTSD
Acronym: DORMI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of response
Sponsor: State University of New York at Buffalo (Other)
Collaborators: The VA Western New York Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ali El Solh, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RF-1070471
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-10

CONDITIONS: Insomnia
Keywords: sleep apnea, PTSD
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes; Stress Disorders, Post-Traumatic | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ramelteon (Active Comparator): Ramelteon 8 mg po at bedtime
  Interventions: Drug: Ramelteon
- Usual care (Placebo Comparator): education brochure about sleep hygiene
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Ramelteon — 8 mg once daily administered within 30 minutes of bedtime
  Other Names: Rozerem
  Arms: Ramelteon
Other: Usual Care — education brochure about sleep hygiene
  Arms: Usual care

SUMMARY:
Obstructive sleep apnea is commonly reported in Veterans with post-traumatic stress disorder, which can potentiate symptoms of anxiety and depression, daytime symptoms and worsen nightmares. Continuous positive airway pressure is the most effective therapy but adherence to treatment is suboptimal. The overarching theme of the proposal is to compare usual care to Ramelteon, in a randomized, clinical trial, investigating the effectiveness of physiological versus pharmacological intervention on sleep quality of life, insomnia severity and CPAP adherence.

DETAILED DESCRIPTION:
Despite the overall improvement in PTSD symptomatology with CPAP therapy, adherence to CPAP is far worse in Veterans with PTSD (41%) compared to the general population with OSA (70%). Among the factors associated with CPAP non-adherence is the coexistence of insomnia. Complex insomnia defined as the coexistence of comorbid insomnia ans OSA is a frequent diagnosis in military personnel with combat exposure. Similar to prior reports of patients with OSA without PTSD, comorbid insomnia can create a barrier to CPAP therapy. Ramelteon (TAK-375), approved by the Food and Drug Administration for the treatment of insomnia with sleep onset abnormalities, is a neurohormone that functions as a melatonin receptor agonist targeting the MT1 and MT2 receptors located in the suprachiasmatic nucleus of the hypothalamus which regulates the circadian rhythm of the 24-hour sleep-wake cycle.The goal is to test the hypothesis that the administration of insomnia therapy-ramelteon- significantly improves treatment outcomes in Veterans with PTSD and complex insomnia compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤70 years old
* Diagnosis of PTSD as determined by the intake conducted through the PTSD Clinic or the Mental Health Clinic
* Documented obstructive sleep apnea by polysomnography (AHI≥5 or more/hour)
* CPAP non adherence defined as less than 70% of nights with >4h CPAP use despite addressing modifiable barriers for CPAP adherence
* Psychotherapeutic treatment stable for at least 4 weeks prior to randomization
* Capable of giving informed consent

Exclusion Criteria:

* Medical:

  * Acute or unstable chronic medical illness
  * History of narcolepsy and/or cataplexy Use of any of these medications: Fluvoxamine, fluconazole (Diflucan), itraconazole (Sporanox), and ketoconazole (Nizoral); cimetidine (Tagamet); clarithromycin (Biaxin); fluoroquinolones including ciprofloxacin, levofloxacin (Levaquin), moxifloxacin (Avelox), norfloxacin (Noroxin), ofloxacin (Floxin), others; HIV protease inhibitors including indinavir (Crixivan), nelfinavir (Viracept), and ritonavir (Norvir, in Kaletra); nefazodone; rifampin
  * Treatment for seizure disorders
  * Pregnant or lactating
  * History of clinically significant hepatic impairment
  * History of hypersensitivity, intolerance, or contraindication to ramelteon
  * Unwilling to try or use CPAP

Psychiatric/Behavioral:

* Diagnosis of current schizophrenia or schizoaffective disorder
* Diagnosis of a substance dependence/abuse disorder in the past year
* Severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to patient or others
* Diagnosis of bipolar disorder
* Consumption of more than two alcoholic beverages per night
* Receiving behavioral or pharmacological treatment for insomnia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 12 weeks post randomization
  Quality of life

SECONDARY OUTCOMES:
PCL-5 | 12 weeks post randomization
  PTSD Checklist
ISI | 12 weeks post randomization
  Insomnia Severity Index
CPAP adherence | 12 weeks post randomization
  CPAP adherence

CONTACTS AND LOCATIONS:
Overall Officials: Ali El Solh, MD, Principal Investigator — The VA Western New York
Locations (1):
- Veterans Affairs Medical Center in Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided